CLINICAL TRIAL: NCT01553916
Title: Phase I/II Trial of Lithium as a Neuroprotective Agent for Patients With Small Cell Lung Cancer (SCLC) Treated With Prophylactic Cranial Irradiation (PCI)
Brief Title: Neuroprotective Effects of Lithium in Patients With Small Cell Lung Cancer Undergoing Radiation Therapy to the Brain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201202073
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Lithium Carbonate; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Lithium carbonate + prophylactic cranial irradiation (Experimental): Lithium carbonate 300 mg PO BID for 7 days prior to the start of prophylactic cranial irradiation (PCI) and will be continued during PCI.
  PCI will be given at 2.5 Gy per fraction, 5 days per week, for 2 weeks to a total dose of 25 Gy, starting on Day 8 after 7 days of lithium.
  Interventions: Drug: Lithium Carbonate; Radiation: Prophylactic cranial irradiation

INTERVENTIONS:
Drug: Lithium Carbonate
  Other Names: Eskalith, Lithane, Lithium, Lithobid, Lithonate, Lithotabs
Radiation: Prophylactic cranial irradiation
  Other Names: PCI

SUMMARY:
This phase I/II trial studies the effects and safety of giving lithium carbonate (lithium) to patients with small cell lung cancer (SCLC) undergoing radiation therapy to the brain (PCI; prophylactic cranial irradiation). PCI is used to prevent cancer metastases from returning in the brain. This treatment can cause short-term memory problems by damaging the hippocampus. Lithium may help prevent or lessen memory problems caused by PCI by protecting the hippocampus.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed small cell lung cancer. Patients with either limited or extensive stage disease are eligible.
* Patient must have completed 4-6 cycles of platinum-based chemotherapy (+/- thoracic radiotherapy).
* Patient must have no evidence of progressive disease on restaging imaging within 3 months of enrollment
* For patients taking medications known to have a significant interaction with lithium carbonate, these medications should be discontinued at least 1 week prior to and during lithium treatment
* Patient must be > or = 18 years old.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 3.0 x IULN
* Creatinine within normal institutional limits OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patient must have an electrocardiogram without evidence of arrhythmia, QT prolongation (QTc > 450 ms in males and > 470 ms in females), or other severe dysfunction within 2 weeks of initiation of lithium
* Women of childbearing potential (women with regular menses, women with amenorrhea, women with irregular cycles, women using a contraceptive method that precludes withdrawal bleeding, and women who have had a tubal ligation) are required to have a negative urine pregnancy test within 14 days prior to the first dose of lithium.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately
* Patient (or legally authorized representative if applicable) must be able to understand and willing to sign an Internal Review Board (IRB) approved written informed consent document

Exclusion Criteria:

* Patient must not have history of prior cranial radiotherapy
* Patient must not have brain metastases present prior to initiation of initial therapy or PCI
* Patient must not have evidence of progressive disease
* Patient must not have received chemotherapy within 3 weeks of initiation of PCI
* Patient must not have a history of other malignancy =< 2 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix
* Patient must not be actively receiving any other investigational agents
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to lithium carbonate
* Patient must not have any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient must not have any uncontrolled thyroid disease
* Patient must not have a seizure disorder
* Patient must not be pregnant and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04-26 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washinton University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Started | 19
Completed | 16
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Pre-treatment MRI metastatic disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 58 [49 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Safety of Lithium Carbonate as Measured by Number of Patients in the Safety lead-in Who Experienced a Dose-limiting Toxicity (DLT)
Description: -Graded and described using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4. Safety will be defined as < 2 patients experiencing DLTs of the first 6 treated.
Time Frame: 3 weeks
Population: -Only patients enrolled in the safety lead-in were evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Immediate Recall Memory Deterioration as Measured by the Hopkins Verbal Learning Test - Immediate Recall (HVLT-IR) Total Score
Description: * The HVLT is a word learning test measuring episodic visual memory
  * The immediate recall memory deterioration test portion consists of 36 words split into 3 sections (animals, gemstones, places of shelter, types of birds, tools, items of clothing, kitchen utensils,weapons, and alcoholic beverages)
  * The words were read aloud and the participants was asked to freely recall them immediately. The list was read a second time followed by a second free recall trial. This was followed by a third reading and third free recall.
  * The words recalled for each trial were recorded and a total recall score tallied (range: 0-36).
  * The higher the score the better the recall
Time Frame: 3 months
Population: 6 participants were not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 13
scores on a scale | 20.0714 (8.29703)

3. Secondary Outcome: Immediate Recall Memory Deterioration as Measured by the Hopkins Verbal Learning Test - Immediate Recall (HVLT-IR) Total Score
Description: as for outcome 2
Time Frame: 6 months
Population: 11 participants were not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 8
scores on a scale | 20.2 (7.22342)

4. Secondary Outcome: Immediate Recall Memory Deterioration as Measured by the Hopkins Verbal Learning Test - Immediate Recall (HVLT-IR) Total Score
Description: as for outcome 2
Time Frame: 12 months
Population: 13 participants were not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 6
scores on a scale | 24.0 (4.89898)

5. Secondary Outcome: Delayed Recall Memory Deterioration as Measured by the Hopkins Verbal Learning Test - Delayed Recall (HVLT-DR) Total Score
Description: * The HVLT is a word learning test measuring episodic visual memory
  * The delayed recall memory deterioration test portion consists of 36 words split into 3 sections (animals, gemstones, places of shelter, types of birds, tools, items of clothing, kitchen utensils,weapons, and alcoholic beverages)
  * The words were read aloud and the participants was asked to freely recall them 20-25 minutes later.
  * The words recalled were recorded and a total recall score tallied (range: 0-36).
  * The higher the score the better the recall
Time Frame: 3 months
Population: -8 participants were not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 11
scores on a scale | 8.6923 (2.89783)

6. Secondary Outcome: Delayed Recall Memory Deterioration as Measured by the Hopkins Verbal Learning Test - Delayed Recall (HVLT-DR) Total Score
Description: as for outcome 5
Time Frame: 6 months
Population: 11 participants were not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 8
scores on a scale | 10.3 (1.56702)

7. Secondary Outcome: Delayed Recall Memory Deterioration as Measured by the Hopkins Verbal Learning Test - Delayed Recall (HVLT-DR) Total Score
Description: as for outcome 5
Time Frame: 12 months
Population: 13 participants were not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 6
scores on a scale | 10.5 (0.83666)

8. Secondary Outcome: Changes in Quality-of-life as Measured by Overall Quality of Life Using the EORTC QLQ30
Description: * Assessed by comparing questionnaire test scores to baseline; European Organization for Research and Treatment of Cancer (EORTC) QLQ30 (global health/QOL, cognitive functioning, and fatigue scales)
  * 30 total questions with 28 questions having answers ranging from 1-4 with 1=not at all and 4= very much and 2 questions ranging from 0-7 with 1-very poor and 7=excellent
  * Raw scores will be transformed to a 100-point scale (0=lowest score, 100=highest score)
  * The higher the score the lower the quality of life
Time Frame: 3 months
Population: 5 participants were not analyzed for this outcome measure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 14
scores on a scale | 45.0820 (7.4469)

9. Secondary Outcome: Changes in Quality-of-life as Measured by Overall Quality of Life Using the Total Score of the EORTC QLQ-BN20
Description: Assessed by comparing questionnaire test scores to baseline; BN20 (future uncertainty and communications deficit scales)
  * 20 questions with answers ranging from 1-4 with 1=not at all and 4=very much
  * Raw scores will be transformed to a 100-point scale (0=lowest score, 100=highest score)
  * The higher the score the lower quality of life
Time Frame: 12 months
Population: 5 participants were not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 14
scores on a scale | 20.5514 (13.8067)

10. Secondary Outcome: Feasibility of Performing Serial Neurocognitive Testing and Quality of Life Exams as Measured by Number of Patients Who Complete the Neurocognitive Testing and Quality of Life Exams
Description: -Defined as at least 4 of 6 patients successfully completing pre-treatment and 3 month post-treatment testing
Time Frame: 3 months
Population: (1) participant is not evaluable as the participant did not start treatment due to pre-treatment MRI showing metastatic disease in spine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 18
Participants | 13

11. Secondary Outcome: Change in Hippocampal Morphology Following Lithium + PCI as Measured by Total Hippocampal Volume
Time Frame: Baseline through 12 months
Population: * 10 participants were evaluable for this outcome measure
  * Originally the outcome measure time frame was baseline through 12 months but there was insufficient data to statistically analyze the change in hippocampal morphology at 12 months due to the number of participants still alive for the 12 month scan.
Measure: Median (Full Range); unit: cc
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 10
cc
  Baseline | 6.13 [5.63 to 7.65]
  3 months | 6.08 [4.95 to 6.69]
  12 months: number analyzed (Participants) | 5
  12 months | 6.34 [5.2 to 6.8]

12. Secondary Outcome: Number of Participants With Brain Metastases
Description: 1-year rate of brain metastases
Time Frame: 12 months
Population: 7 participants were not evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 9
Participants | 2

13. Secondary Outcome: Number of Central Nervous System (CNS) Adverse Events
Description: Adverse events will be tabulated by type and grade using NCI CTCAE v 4.
Time Frame: Through 12 months
Measure: Number; unit: CNS adverse events
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 19
CNS adverse events
  Grade 1 | 28
  Grade 2 | 6
  Grade 3 | 2

14. Secondary Outcome: Rate of Overall Survival
Description: -Overall survival is defined as the time between date of on study and date of death due to any cause
Time Frame: 12 months
Population: 7 participants were not evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Number analyzed (Participants) | 9
Participants | 5

ADVERSE EVENTS:
Arm/Group | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Lithium Carbonate + Prophylactic Cranial Irradiation (N=19)
Anemia (Blood and lymphatic system disorders) | 6
Red blood cell decrease (Blood and lymphatic system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 2
Floaters (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 2
Edema face (General disorders) | 1
Fatigue (General disorders) | 11
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 2
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Bronchial infection (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Creatinine increased (Investigations) | 2
INR increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Weight gain (Investigations) | 1
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 7
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Other - sacroiliac pain (Musculoskeletal and connective tissue disorders) | 1
Other - right leg pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Other - disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 10
Memory impairment (Nervous system disorders) | 2
Nystagmus (Nervous system disorders) | 1
Other - myoclonic jerk (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes